CLINICAL TRIAL: NCT02300987
Title: A Randomized, Blinded, Placebo-controlled, Phase II Trial of LEE011 in Patients With Relapsed, Refractory, Incurable Teratoma With Recent Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLEE011X2201; 2014-000428-12 (EudraCT Number)
Record Dates: First submitted 2014-07-15; First posted 2014-11-25 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Teratoma
Keywords: Teratoma,; Germ Cell tumor,; incurable teratoma,; CDK4/6,; LEE011
MeSH Terms: conditions — Teratoma; Neoplasms, Germ Cell and Embryonal | interventions — ribociclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LEE011 (Active Comparator): 600 mg daily dosing days 1-21 of a 28 day cycle
  Interventions: Drug: LEE011
- Placebo Arm (Placebo Comparator): 600 mg daily dosing days 1-21 of a 28 day cycle
  Interventions: Drug: LEE011 Placebo

INTERVENTIONS:
Drug: LEE011
  Arms: LEE011
Drug: LEE011 Placebo
  Arms: Placebo Arm

SUMMARY:
This was a multi-center, randomized, double blind (investigator and subject), placebo controlled Phase II study to determine the efficacy and safety of treatment with ribociclib versus placebo in subjects with progressive relapsed, refractory incurable teratoma. Eligible subjects were randomized in a 2:1 ratio to ribociclib or placebo.

After discontinuation of study treatment, patients were followed up for safety, disease progression and overall survival.

DETAILED DESCRIPTION:
Safety follow-up: After discontinuation of study treatment, all subjects were followed for safety for 30 days except in the case of death, loss to follow up, withdrawal of consent, or discontinuation of study treatment to enroll in the ribociclib rollover clinical trial (CLEE011X2X01B).

Disease progression follow-up: Subjects who discontinued study drug for any reasons other than disease progression were followed for efficacy every 8 weeks during the first 12 months. After 12 months, they were followed for every 12 weeks until disease progression, death, discontinuation from the study for any other reason (i.e. loss to follow-up or withdrawal of consent), the initiation of a new antineoplastic treatment, or until all subjects had been followed for at least 18 months after their first dose of study drug, or early study termination, whichever occurred first.

Survival follow-up: All subjects were followed for survival via a phone call (or during a clinic visit) every 12 weeks and up to one additional time per quarter if a survival update was required to meet safety or regulatory needs. The safety follow-up was carried out until any of the following occurred (whichever occurred first): death, withdrawal of consent, loss to follow-up, at least 18 months had elapsed from when the last subject had started treatment, or when 80% of subjects had died or were lost to follow-up, or early study termination.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of teratoma for which no additional standard surgical or medical therapy exists
* Patients must have completed at least 1 prior line of chemotherapy for germ cell tumor (except patients who present with primary pure teratoma who need not have received any previous chemotherapy)
* Radiographic progression, defined by RECIST v.1.1, after the last cancer treatment and within 12 weeks prior to enrollment, compared with scans within 1 year of enrollment.
* Availability of an archival or newly obtained tumor sample (collected at diagnosis or progression) with accompanying pathology report
* Meaurable or evaluable extra-cranial disease as defined by RECIST v 1.1

Key Exclusion Criteria:

* Malignant germ cell tumors with mixed histology such as embryonal carcinoma, choriocarcinoma, yolk sac tumor or seminoma. Note - this refers to the histology at the time of enrollment, not the histolgy at the time of initial presentation.
* Pathologic evidence of malignant transformation
* CNS disease unless radiation therapy and/or surgery has been completed and serial evaluation demonstrates stable disease
* Prior treatment with any CDK4/6 inhibitor therapy
* Systemic antineoplastic therapy or any experimental therapy within 3 weeks before the first dose of study drug (6 weeks for prior nitrosoureas, bevacizumab, or mitomycin C)
* Major surgery ≤ 2 weeks or radiotherapy ≤ 4 weeks prior to planned start of study drug or patient has not recovered from major side effects.
* Requirement for treatment with any of the prohibited medications including strong CYP3A inhibitors, strong CYP3A inducers, CYP3A substrates with a narrow therapeutic index, and medications with strong risk of QT prolongation

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (3):
  - USC Kenneth Norris Comprehensive Cancer Center Oncology Dept, Los Angeles, California
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Memorial Sloan Kettering Oncology Department., New York, New York
- Novartis Investigative Site, Villejuif, France
- Novartis Investigative Site, Groningen, Netherlands
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomly assigned to Ribociclib or Placebo in a 2:1 ratio. The 2 subjects from the placebo group (primary phase) entered the secondary treatment phase (cross over) after they experienced disease progression, and were then treated with LEE01. One patient from the LEE arm entered the secondary treatment phase.
Pre-assignment Details: 42 subjects were planned to be included (28 for the LEE011 arm and 14 for the Placebo arm). The study was stopped prematurely with 10 patients randomized and treated in this study (8 in the ribociclib arm, 2 in the placebo arm).
Period: Primary Phase : Prior to Cross-over
Arm/Group | LEE011 | Placebo Arm
Started | 8 | 2
Completed | 2 | 0
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — progressive disease | 3 | 2
Period: Secondary Phase : Cross-over to LEE011
Arm/Group | LEE011 | Placebo Arm
Started | 1 | 2
Completed | 0 | 1
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEE011 | Placebo Arm | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: full analysis set
  years | 32.3 (6.76) | 40.5 (17.68) | 33.9 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Ful analysis set
  Participants
    Female | 0 | 0 | 0
    Male | 8 | 2 | 10
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full analysis set
  Participants
    Caucasian | 4 | 1 | 5
    Native American | 1 | 0 | 1
    Unknown | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Date of randomization to the date of the first documented progression or death due to any causeas per RECIST v1.1 (by local investigator assessment). Only includes data prior to cross over. Disease progression follow-up: Subjects who discontinued study drug for any reasons other than disease progression were followed for efficacy every 8 weeks during the first 12 months. After 12 months, they were followed for every 12 weeks until disease progression, death, discontinuation from the study for any other reason (i.e. loss to follow-up or withdrawal of consent), the initiation of a new antineoplastic treatment, or until all subjects had been followed for at least 18 months after their first dose of study drug, or early study termination, whichever occurred first.
Time Frame: At 24 months
Population: Full analysis set. After 10 subjects were enrolled and treated, the recruitment was halted due to business reasons.There were no safety concerns which contributed to the decision to halt enrollment. Limited efficacy analyses were performed.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
Days | 71.4 [33.9 to 90.1] | 0.0 [0.0 to 0.0]

2. Secondary Outcome: Best Overall Response (BOR)
Description: as per RECIST v1.1. Only includes data prior to cross over. Placebo arm : the subject who experienced SD as best overall response entered the secondary phase and was treated with LEE011 after he experienced progressive disease, following his best Stable Disease response. In this outcome measure 2, only the best overall response is indicated.
Time Frame: At 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
Participants
  Stable Disease (SD) | 8 | 1
  Progressive Disease (PD) | 0 | 1

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) = complete response (CR) or partial response (PR).
  ORR was zero, as there were no CRs or PRs in either of the groups
Time Frame: At 27 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
percentage of participants | 0 [0.0 to 36.9] | 0 [0.0 to 84.2]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: as per RECIST v1.1. Only includes data prior to cross over. Placebo arm : the disease control rate is based on the best overall response described in the outcome measure 2.
Time Frame: At 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
percentage of participants | 100 [63.1 to 100.0] | 50 [1.3 to 98.7]

5. Secondary Outcome: Overall Survival (OS)
Description: Only includes data prior to cross over. OS defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut off, OS was censored at the date of last known date patient alive
Time Frame: At 27 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
Participants | 6 [27.6 to 92.5] | 1 [0.6 to 91.0]

6. Secondary Outcome: Overall Survival Rate
Description: as per RECIST v1.1. Only includes data prior to cross over. Kaplan-Meier estimates (%) OS rate [95% CI] at different timepoints. The overall survival rate at 27 month is 72.9% by Kaplan-Meyer (K-M) estimator; the reason that it is not 75% (1-25%) (Overall survival) is because of censoring. When the other 6 patients were censored would impact the survival rate with K-M method as the number of patients at risk after each censor was changed.
  NA for the 95% CI is indicated when no patient died at the time of assessment, as the CI could not be calculated as per definition. Results are presented as a % calculated on the total number of participants.
Time Frame: 1, 2, 3, 6, 9, 12, 15, 18, 21, 24 and 27 months
Population: Full analysis set.After 10 subjects were enrolled and treated, the recruitment was halted due to business reasons.There were no safety concerns which contributed to the decision to halt enrollment. Limited efficacy analyses were performed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
Percentage of Participants
  1 month | 100 [NA to NA] — NA represents not estimable. | 100 [NA to NA] — NA represents not estimable.
  2 months | 100 [NA to NA] — NA represents not estimable. | 100 [NA to NA] — NA represents not estimable.
  3 months | 100 [NA to NA] — NA represents not estimable. | 100 [NA to NA] — NA represents not estimable.
  6 months | 100 [NA to NA] — NA represents not estimable. | 100 [NA to NA] — NA represents not estimable.
  9 months | 100 [NA to NA] — NA represents not estimable. | 100 [NA to NA] — NA represents not estimable.
  12 months | 87.5 [38.7 to 98.1] | 100 [NA to NA] — NA represents not estimable.
  15 months | 87.5 [38.7 to 98.1] | 100 [NA to NA] — NA represents not estimable.
  18 months | 87.5 [38.7 to 98.1] | 100 [NA to NA] — NA represents not estimable.
  21 months | 87.5 [38.7 to 98.1] | 50.0 [0.6 to 91.0]
  24 months | 87.5 [38.7 to 98.1] | 50.0 [0.6 to 91.0]
  27 months | 72.9 [27.6 to 92.5] | 50.0 [0.6 to 91.0]

7. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths are collected from first patient first visit up to 30 days after study treatment discontinuation (approximately 12 months, median duration of exposure). Patients with cancer are also followed up for overall survival until the end of the trial. During overall survival (up to 27 months after the first patient first visit), additional deaths were recorded, including deaths due to the cancer disease (having occurred more than 30 days after study drug discontinuation)
Time Frame: 12 months, 27 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEE011 | Placebo Arm
Number analyzed (Participants) | 8 | 2
Participants
  Total deaths | 2 | 1
  Deaths on treatment | 0 | 0
  Deaths post treatment survival follow up | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, as defined in the study protocol, for a median duration of exposure of 385 days.
Description: Any sign or symptom that occurs during the study treatment and 30 days post treatment follow up.
Groups:
- Placebo: Placebo
- All Patients: All patients
Arm/Group | LEE011 | Placebo | All Patients
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/2 | 3/10
Other Adverse Events (participants affected / at risk) | 8/8 | 1/2 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEE011 (N=8) | Placebo (N=2) | All Patients (N=10)
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEE011 (N=8) | Placebo (N=2) | All Patients (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 0 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3
Asthenia (General disorders) | 3 | 0 | 3
Breakthrough pain (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 3
Impaired healing (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 2
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 0 | 3
Anal infection (Infections and infestations) | 1 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alpha 1 foetoprotein increased (Investigations) | 1 | 0 | 1
Blood creatine increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 2
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 6 | 0 | 6
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0 | 3
Libido decreased (Psychiatric disorders) | 1 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
After 10 patients were included the recruitment was halted for business reasons not for safety concerns. Overall Survival presents all deaths up to 27 months while the all-cause mortality presents deaths up to 30 days after treatment discontinuation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis'agreements with its investigators may vary. However Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT02300987/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT02300987/SAP_001.pdf